CLINICAL TRIAL: NCT01767558
Title: Phased RF Evaluation of Acute Pulmonary Vein Isolation in Paroxysmal AF With New GENius UI and PVAC GOLD
Brief Title: PRECISION GOLD Post Market Study in Europe of Pulmonary Vein Ablation Catheter (PVAC GOLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRECISION GOLD
Record Dates: First submitted 2013-01-08; First posted 2013-01-14 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ablation / MRI (Other): All subjects will undergo a standard of care ablation procedure for paroxysmal AF with the CE-Marked PVAC GOLD catheter.
  MRIs will be performed on all subjects at Enrollment and Pre-Discharge (Post Ablation). Subjects with a positive MRI (cerebral lesion) at Pre-Discharge will undergo another MRI at the 1 month follow-up visit.
  Interventions: Other: Ablation / MRI

INTERVENTIONS:
Other: Ablation / MRI — All subjects will undergo a standard of care ablation procedure for paroxysmal AF with the CE-Marked PVAC GOLD catheter.
  MRIs will be performed on all subjects at Enrollment and Pre-Discharge (Post Ablation). Subjects with a positive MRI (cerebral lesion) at Pre-Discharge will undergo another MRI at the 1 month follow-up visit.

SUMMARY:
PRECISION GOLD is a prospective, multi-center, single arm, unblinded interventional post market clinical study conducted in Europe. The purpose of the study is to evaluate asymptomatic cerebral embolic (ACE) lesions in subjects with symptomatic paroxysmal atrial fibrillation undergoing ablation with the Pulmonary Vein Ablation Catheter (PVAC) GOLD.

DETAILED DESCRIPTION:
10-12 centers in Europe will enroll up to 56 subjects who meet the inclusion/exclusion criteria and provide consent to participate in the study. Subjects will undergo an ablation for paroxysmal AF with the Medtronic PVAC GOLD (CE-Mark). To assess for ACE lesions, pre- and post-ablation procedure cerebral MRIs will be done along with a neurological exam (Mini Mental State Exam). Subjects will be followed for 1 month post-procedure when a repeat MRI and neurological exam will be conducted if the subject had a positive MRI at pre-hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic AF (>/=2 recurrent AF episodes that self terminate or AF </=48 hours that are cardioverted)
* Documentation of >/=1 paroxysmal AF events within past year
* AF symptoms (e.g. palpitations, fatigue, exertional dyspnea, effort intolerance)
* Prescribed to vitamin K antagonist (e.g. warfarin/coumadin)
* Age 18-70 years old
* Clinically indicated for a pulmonary vein ablation
* Willing and able to give informed consent
* Willing, able and committed to participate in all study required activities for the duration of the study

Exclusion Criteria:

* Diagnosis of persistent or permanent AF
* Prior left atrial ablation
* Presence of intracardiac thrombus
* Contraindicated for vitamin K antagonist
* Prescribed to direct thrombin or factor inhibitors (e.g. dabigatran, rivaroxaban)
* Prescribed to any investigational drug that may confound the study results
* Cardiac valve prosthesis
* Significant congenital heart defect (corrected or not)
* Pulmonary vein stents
* Pre-existing pulmonary vein stenosis
* Cerebral ischemic event (e.g. stroke, TIA) that occurred within 6 months of study consent date
* If female - pregnancy
* Participation in any other cardiovascular clinical study
* Contraindicated for MRI
* Active sepsis
* Blood clotting abnormalities (genetic)
* Presence of left atrial myxoma
* Venous filtering device (e.g. Greenfield filter)
* Invasive cardiac procedure in past 90 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Measure rate of post-procedure asymptomatic cerebral embolic (ACE) as determined by MRI | 1-45 days post-ablation procedure
  Pre- and post-ablation MRIs will be evaluated for ACE lesions. If the post-ablation MRI (within 16-72 hours) is positive for ACE, a repeat MRI will be completed at the 1 month visit.

SECONDARY OUTCOMES:
Measure acute procedural success | 0-1 days after procedure
  Acute procedural success is defined as:
  * Only PVAC GOLD catheters used to achieve pulmonary vein (PV) isolation
  * All accessible PVs were isolated (entrance block)
  * Sinus rhythm is restored at the end of the ablation procedure (with or without cardioversion)
Report procedure and/or device related serious adverse events using PVAC GOLD | 0-45 days post-ablation procedure

CONTACTS AND LOCATIONS:
Locations (11):
- ZNA Middelheim, Antwerp, Belgium
- Hopital Cardiolgique du Haut-Leveque, Pessac, France
- Germany (3):
  - Zentraklinik Bad Berka, Bad Berka
  - St. Agnes Hospital Bocholt, Bocholt
  - Zentrum fuer klinische Pruefungen in der Facharztzentrum Dresden-Neustadt GbR, Dresden
- Debrecen University, Debrecen, Hungary
- Netherlands (2):
  - Catharina Hospital, Eindhoven
  - St. Antonius Hospital, Nieuwegein
- United Kingdom (3):
  - Eastbourne District General Hospital, Eastbourne
  - University Hospital of South Manchester, Manchester
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] De Greef Y, Dekker L, Boersma L, Murray S, Wieczorek M, Spitzer SG, Davidson N, Furniss S, Hocini M, Geller JC, Csanadi Z; PRECISION GOLD investigators. Low rate of asymptomatic cerebral embolism and improved procedural efficiency with the novel pulmonary vein ablation catheter GOLD: results of the PRECISION GOLD trial. Europace. 2016 May;18(5):687-95. doi: 10.1093/europace/euv385. Epub 2016 Jan 29. PMID 26826134